CLINICAL TRIAL: NCT00997256
Title: Phase I, Placebo-controlled, Double-blind, Randomised, Single-centre Study of Single Cross-over Design to Investigate the Effects of the Herbal Preparation Neurapas® Balance Compared With Placebo on Sleep EEG, Mental Performance and Well-being
Brief Title: Study to Investigate Effects of a Herbal Drug Compared to Placebo on Sleep
Acronym: sleep-EEG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pascoe Pharmazeutische Praeparate GmbH (Industry)
Responsible Party: Anja Braschoss, Pascoe Pharmazeutische Preparate GmbH
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSC 152/04
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Last update posted 2010-05-17 (Estimated); Status verified 2010-05

CONDITIONS: Healthy; Sleep Quality
Keywords: sleep-EEG; sleep architecture; sleep duration; sleep continuity; REM-sleep; vigilance; well-being; Healthy volunteers
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Valeriana extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Verum (Experimental): Neurapas balance, film-coated tablets
  Interventions: Drug: Neurapas® balance (Herbal product (Hypericum, Passionflower, Valerian))
- Placebo (Placebo Comparator): Film-coated sugar-pill
  Interventions: Drug: film-coated sugar-pill

INTERVENTIONS:
Drug: Neurapas® balance (Herbal product (Hypericum, Passionflower, Valerian)) — 3 x 2 tablets / day over 3 days
  Other Names: Neurapas balance, film-coated tablet over 3 days
  Arms: Verum
Drug: film-coated sugar-pill — 3 x 2 tablets / day over 3 days
  Arms: Placebo

SUMMARY:
To demonstrate the influence of a herbal preparation containing hypericum, passionflower, and valerian on sleep structure, improvement of attention, and well-being in comparison to placebo.

DETAILED DESCRIPTION:
To demonstrate the influence of the herbal combination preparation Neurapas® balance on the objective sleep structure in comparison with placebo. A further aim was to investigate whether treatment with Neurapas® balance versus placebo brings about an improvement in attention and well-being and whether these changes are related to the improvement in the sleep structure.

1. Does the administration of 3 x 2 Neurapas® balance tablets over a period of three days vs. placebo lead to an improvement in continuity of sleep?
2. Does the administration of 3 x 2 Neurapas® balance tablets over a period of three days vs. placebo lead to an improvement in sleep architecture, especially an increase in deep sleep?
3. Does the administration of 3 x 2 Neurapas® balance tablets over a period of three days vs. placebo lead to an improvement in morning attentional performance?
4. Does the administration of 3 x 2 Neurapas® balance tablets over a period of three days vs. placebo lead to an improvement in morning well-being?

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged between 18 and 55 years
* Normal sleeping times (at least 6 hours a night), going to sleep between 22.00 and 1.00 hours, getting up between 6.00 and 9.00 hours
* Written informed consent
* The volunteer is willing and able to cooperate fully
* The volunteer agrees not to drink any alcohol for the duration of the study

Exclusion Criteria:

* Participation in another study in the last 30 days or participation in this study at an earlier date
* Lack of verbal or intellectual ability to communicate adequately and to understand the information to volunteers
* Legal incompetence
* Smoker
* Shift worker
* Transatlantic flight in the last 4 weeks
* Taking psychotropic drugs within the last 4 weeks
* Taking medicines that influence the EEG within the last 4 weeks
* Diseases that influence the sleep EEG
* History of known medication / drug / alcohol misuse according to ICD-10 coding F10 - F19
* Known intolerance/hypersensitivity/allergy to St. John's wort, valerian or passionflower
* Taking inadmissible concomitant medication (anxiolytic, neuroleptic or hypnotic drugs, cyclosporin, sedative, sleep-promoting or mood-enhancing medicines, antidepressants other than the trial medication, coumarin-type anticoagulants, oral contraceptives, tranquillisers, homeopathic remedies, digoxin, theophylline, indinavir, nortriptyline, amitriptyline)
* Known light-sensitivity

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2004-12; Primary Completion 2005-01 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of sleep by Polysomnography (sleep continuity and sleep architecture) | Day 3 + 14

SECONDARY OUTCOMES:
Attention Stress Test d2 (Brickenkamp) | Day 4 + 15
Alertness and vigilance test (TAP) | Day 4 + 15
Trail-Making Test (TMT) | Day 4 + 15
Questionnaire on physical symptoms of subjective well-Being(MKSL, Janke) | Day 4 +15
Questionnaire on psychological aspects of well-being(BSKE, Janke) | Day 4 + 15
ZERSSEN Scale of evaluation of subjective well-being (Bf-S) | Day 4 + 15
Sleep Questionnaire(SF) | Day 4 + 15

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich M Hemmeter, PD Dr Dr, Principal Investigator — Phillipps University Marburg, Clinic for Psychiatry and Psychotherapy
Locations (1):
- Phillipps University, Clinic for Psychiatry and Psychotherapy, Marburg, Hesse, Germany